CLINICAL TRIAL: NCT02193958
Title: A Phase 1/2a, Dose Escalation Study of FF-10501-01 for the Treatment of Advanced Hematologic Malignancies
Brief Title: Study of FF-10501-01 in Patients With Relapsed or Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF1050101US01
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: AML; CMML; MDS
Keywords: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Phase 1 Cohort 1: 50mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 2: 100mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 3: 200mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 4: 300mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 5: 400mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 6: 500mg/m2 (Experimental): FF-10501-01 tablets BID every 14 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 2a Cohort 7: 400mg/m2 in MDS/CMML (Experimental): FF-10501-01 tablets BID every 21 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01
- Phase 1 Cohort 8: 400mg/m2 (Experimental): FF-10501-01 tablets BID every 28 days of a 28 day cycle.
  Interventions: Drug: FF-10501-01
- Phase 2a Cohort 9: 400mg/m2 (Experimental): FF-10501-01 tablets BID every 21 days of a 28-day cycle.
  Interventions: Drug: FF-10501-01

INTERVENTIONS:
Drug: FF-10501-01 — FF-10501-01 will be administered orally on Days 1-14 of a 28-day cycle (Cohorts 1-6), Days 1-21 of a 28-say cycle (Cohort 7), Days 1-28 of a 28-day cycle (Cohort 8) or Days 1-21 of a 28-say cycle (Cohort 9). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Other Names: Single Group Assignment; Drug FF-10501-01

SUMMARY:
A Phase 1/2a Dose Escalation Study of FF-10501-01 in Patients with Relapsed or Refractory Hematological Malignancies to determine the safety and tolerability. A total of 6 cohorts will be enrolled in Phase 1 to establish the MTD. A total of 20 subjects with MDS/CMML treated at the RP2D are planned, including MDS/CMML subjects treated at the RP2D in Phase 1.

DETAILED DESCRIPTION:
Subjects will receive FF-10501-01 orally on a twice daily schedule for 14, 21 or 28 days repeated every 28 days (=1 cycle). Disease assessments, including analysis of blood and bone marrow aspirates, will be performed at the end of Cycle 1 and every 2 cycles thereafter. Subjects who demonstrate objective response or stable disease will be allowed to continue therapy with FF-10501-01 until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in condition that prevent further study participation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced hematologic malignancies;

Phase 1:

* High-risk MDS/CMML (defined as ≥ 10% peripheral blood or marrow blasts and/or IPSS score ≥ 1.5) and relapsed or refractory to prior therapy
* AML relapsed or refractory to prior therapy, or ≥ 60 years of age and not a candidate for other therapies

Phase 2a:

* MDS/CMML, relapsed from, or refractory to, prior HMA therapy; the latter defined as failure to achieve clinical remission (CR), partial remission (PR) or hematologic improvement (HI) after previous HMA therapy (≥ 4 cycles of azacitidine or decitabine), or progression during, or toxicity to previous HMA therapy precluding further HMA treatment, and,
* Bone marrow blast count ≥ 10% or peripheral blast count ≥ 5%, or IPSS-R score ≥ 3.5.

  * At least 3 weeks beyond the last chemotherapy, targeted anticancer agent, major surgery or experimental treatment and recovered from all acute toxicities (≤ Grade 1). Hydroxyurea used to control peripheral blast counts is permitted up to Day 7 of treatment on study.
  * Adequate performance status: ECOG ≤ 2;
  * Adequate renal and hepatic function:
* creatinine ≤ 2.0 mg/dL, or calculated creatinine clearance ≥ 45 mL/min
* total bilirubin ≤ 2 times the upper limit of normal (ULN)
* ALT/AST ≤ 2 times ULN

  * Negative serum pregnancy test
  * Ability to provide written informed consent

Exclusion Criteria:

* Known history of coronary artery disease, angina, myocardial infarction, congestive heart failure, cardiac arrhythmia or any other type of heart disease present within the last 6 months
* Known family history of hereditary heart disease
* QT interval corrected for rate (QTc) > 450 msec on the electrocardiogram (ECG) obtained at Screening
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, with the exception of anti-microbials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for the care of the patient.
* Presence of active central nervous system (CNS) leukemia. Subjects adequately treated for CNS leukemia documented by 2 consecutive cerebrospinal fluid samples negative for leukemia cells are eligible. Subjects with no history of CNS leukemia will not be required to undergo cerebrospinal fluid sampling for eligibility.
* Known positive for HIV, hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV).
* Active infection requiring IV anti-infective usage within the last 7 days prior to study treatment.
* Any other medical intervention or condition which could compromise adherence to study requirements or confound the interpretation of study results.
* Pregnant or breast-feeding.
* Treatment with any investigational product within 28 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Cleveland Clinic at Taussig Cancer Center, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Manero G, Pemmaraju N, Alvarado Y, Naqvi K, Ravandi F, Jabbour E, De Lumpa R, Kantarjian H, Advani A, Mukherjee S, Gerds A, Carraway HE, Nazha A, Iwamura H, Murase M, Bavisotto L, Kurman M, Maier G, Johansen M, Sekeres MA. Results of a Phase 1/2a dose-escalation study of FF-10501-01, an IMPDH inhibitor, in patients with acute myeloid leukemia or myelodysplastic syndromes. Leuk Lymphoma. 2020 Aug;61(8):1943-1953. doi: 10.1080/10428194.2020.1747065. Epub 2020 Apr 7. PMID 32264726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 2 academic medical centers between July 2014 and December 2018. The first participant was enrolled on August 21, 2014 and the last participant was enrolled on December 3, 2018. Study completion date was August 9, 2019.
Pre-assignment Details: For Phase 1, anticipated enrollment was 48 subjects; 38 subjects were enrolled and treated with FF-10501-01.
  For Phase 2, anticipated enrollment was 20 subjects; 17 were enrolled and treated with FF-10501-01.
Groups:
- Phase 1 Cohort 1: 50mg/m2: FF-10501-01 tablets BID for 14 days of a 28 day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 2: 100mg/m2; Phase 1 Cohort 3: 200mg/m2; Phase 1 Cohort 4: 300mg/m2: FF-10501-01 tablets BID for 14 days of a 28-day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 5: 400mg/m2: FF-10501-01 tablets BID for 14 days of a 28-day cycle
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 6: 500mg/m2: FF-10501-01 tablets BID every 14 days of a 28-day cycle
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 7: 400mg/m2 in MDS/CMML: FF-10501-01 tablets BID for 21 days of a 28 day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-21 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 8: 400mg/m2: FF-10501-01 tablets BID for 28 days of a 28 day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-28 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 2a Cohort 9: 400mg/m2: FF-10501-01 tablets BID for 21 days of a 28-day cycle
  FF-10501-01: FF-10501-01 will be administered orally on Days 1-21 of a 28-day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
Period: Overall Study
Arm/Group | Phase 1 Cohort 1: 50mg/m2 | Phase 1 Cohort 2: 100mg/m2 | Phase 1 Cohort 3: 200mg/m2 | Phase 1 Cohort 4: 300mg/m2 | Phase 1 Cohort 5: 400mg/m2 | Phase 1 Cohort 6: 500mg/m2 | Phase 1 Cohort 7: 400mg/m2 in MDS/CMML | Phase 1 Cohort 8: 400mg/m2 | Phase 2a Cohort 9: 400mg/m2
Started | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17
Treated | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17
Completed | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 6
Not Completed | 2 | 2 | 4 | 4 | 7 | 5 | 3 | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Cohort 1: 50mg/m2; Phase 1 Cohort 2: 100mg/m2: FF-10501-01 tablets BID for 14 days of a 28 day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle (Cohorts 1-6). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 3: 200mg/m2; Phase 1 Cohort 4: 300mg/m2: FF-10501-01 tablets BID for 14 days of a 28-day cycle.
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle (Cohorts 1-6). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 5: 400mg/m2: FF-10501-01 tablets BID for 14 days of a 28-day cycle
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-14 of a 28-day cycle (Cohorts 1-6). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 6: 500mg/m2: FF-10501-01 tablets BID for 14 days of a 28-day cycle.
  FF-10501-01: FF-10501-01 will be administered orally on Days 1-14 of a 28-day cycle (Cohorts 1-6). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 7: 400mg/m2: FF-10501-01 tablets BID every 21 days of a 28 day cycle.
  FF-10501-01: FF-10501-01 will be administered orally on Days 1-21 of a 28-say cycle (Cohort 7). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 1 Cohort 8: 400mg/m2: FF-10501-01 tablets BID for 28 days of a 28-day cycle
  FF-10501-01: FF-10501-01 will be administered orally BID on Days 1-28 of a 28-day cycle (Cohort 8). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Phase 2a Cohort 9: 400mg/m2: FF-10501-01 tablets BID for 21 days of a 28-day cycle. FF-10501-01 will be administered orally BID on Days 1-21 of a 28-day cycle (Cohorts 9). The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1: 50mg/m2 | Phase 1 Cohort 2: 100mg/m2 | Phase 1 Cohort 3: 200mg/m2 | Phase 1 Cohort 4: 300mg/m2 | Phase 1 Cohort 5: 400mg/m2 | Phase 1 Cohort 6: 500mg/m2 | Phase 1 Cohort 7: 400mg/m2 | Phase 1 Cohort 8: 400mg/m2 | Phase 2a Cohort 9: 400mg/m2 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 1 | 8
  >=65 years | 3 | 2 | 1 | 4 | 7 | 4 | 5 | 5 | 16 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.67 (4.04) | 69.00 (11.79) | 66.25 (9.36) | 76.00 (5.35) | 79.00 (5.72) | 71.00 (9.14) | 77.40 (3.78) | 73.29 (9.36) | 73.00 (6.68) | 73.44 (7.355)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 2 | 3 | 2 | 4 | 3 | 21
  Male | 1 | 1 | 2 | 3 | 5 | 2 | 3 | 3 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 5
  Not Hispanic or Latino | 2 | 3 | 3 | 3 | 2 | 4 | 3 | 7 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 4
  White | 3 | 3 | 3 | 4 | 5 | 5 | 4 | 6 | 16 | 49
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17 | 55

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed by Adverse Events
Description: Safety and tolerability assessed by adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicity (DLT), dose reductions, delays or withdrawals due to toxicity
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Phase 1 Cohort 1: 50mg/m2 | Phase 1 Cohort 2: 100mg/m2 | Phase 1 Cohort 3: 200mg/m2 | Phase 1 Cohort 4: 300mg/m2 | Phase 1 Cohort 5: 400mg/m2 | Phase 1 Cohort 6: 500mg/m2 | Phase 1 Cohort 7: 400mg/m2 | Phase 1 Cohort 8: 400mg/m2 | Phase 2a Cohort 9: 400mg/m2
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17
participants
  Any TEAEs | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17
  Any study drug related TEAEs | 3 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 14
  Any serious TEAEs | 2 | 2 | 4 | 3 | 7 | 5 | 4 | 7 | 11
  Grade 3 or 4 TEAEs | 2 | 2 | 4 | 3 | 6 | 3 | 4 | 7 | 15
  Grade 3 or 4 study drug related TEAEs | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 6
  Interruption of study drug due to TEAEs | 0 | 1 | 2 | 2 | 2 | 2 | 3 | 5 | 7
  Death due to TEAEs | 1 | 1 | 2 | 1 | 3 | 2 | 1 | 3 | 0

2. Secondary Outcome: Determination of Objective Response (OR) Rates.
Description: The OR endpoint: proportion of subjects w/ OR as best response (CR, CRi or PR) assessed at the end of Cycles 1 and 3.
  AML: CR - free of all symptoms related to leukemia, absolute neutrophil count > 1.0 x 10^9/L, platelet count ≥ 100 x 10^9/L, normal bone marrow with < 5% blasts no Auer rods; CRi - CR with residual thrombocytopenia (platelet count < 100 x 10^9/L) or residual neutropenia (absolute neutrophil count < 1.0 x 10^9/L); PR - A ≥ 50% decrease in bone marrow blasts to 5 to 25% abnormal.
  MDS or CMML: CR - free of all symptoms related to leukemia, absolute neutrophil count ≥ 1.0 x 10^9/L, platelet count ≥ 100 x 10^9/L, bone marrow ≤ 5% myeloblasts, w/ normal maturation of all cell lines, hemoglobin ≥ 11g/dL, no blasts in the peripheral blood; PR - All CR criteria with ≥50% decrease in bone marrow blasts over pre-treatment (but still > 5%); Marrow CR - In bone marrow, ≤ 5% myeloblasts and decrease by ≥ 50% over pre-treatment.
Time Frame: OR responses were assessed at end of Cycles 1 thru 3. Each cycle was 28 days in length.
Measure: Number; unit: participants
Arm/Group | Phase 1 Cohort 1: 50mg/m2 | Phase 1 Cohort 2: 100mg/m2 | Phase 1 Cohort 3: 200mg/m2 | Phase 1 Cohort 4: 300mg/m2 | Phase 1 Cohort 5: 400mg/m2 | Phase 1 Cohort 6: 500mg/m2 | Phase 1 Cohort 7: 400mg/m2 | Phase 1 Cohort 8: 400mg/m2 | Phase 2a Cohort 9: 400mg/m2
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 5 | 5 | 7 | 17
participants
  Partial Response subjects | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Complete bone marrow remission (mCR) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Each patient was followed from baseline through the treatment period (maximum treatment period up to 31 months) until long-term follow-up was completed (6 mos post end of study) or patient discontinued either by withdrawal, progressive disease or death.
Description: Definitions do not differ from clinicaltrials.gov
Arm/Group | Phase 1 Cohort 1: 50mg/m2 | Phase 1 Cohort 2: 100mg/m2 | Phase 1 Cohort 3: 200mg/m2 | Phase 1 Cohort 4: 300mg/m2 | Phase 1 Cohort 5: 400mg/m2 | Phase 1 Cohort 6: 500mg/m2 | Phase 1 Cohort 7: 400mg/m2 | Phase 1 Cohort 8: 400mg/m2 | Phase 2a Cohort 9: 400mg/m2
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 3/4 | 4/4 | 7/7 | 4/5 | 2/5 | 5/7 | 8/17
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 4/4 | 3/4 | 7/7 | 5/5 | 4/5 | 7/7 | 15/17
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 4/4 | 7/7 | 5/5 | 5/5 | 7/7 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1: 50mg/m2 (N=3) | Phase 1 Cohort 2: 100mg/m2 (N=3) | Phase 1 Cohort 3: 200mg/m2 (N=4) | Phase 1 Cohort 4: 300mg/m2 (N=4) | Phase 1 Cohort 5: 400mg/m2 (N=7) | Phase 1 Cohort 6: 500mg/m2 (N=5) | Phase 1 Cohort 7: 400mg/m2 (N=5) | Phase 1 Cohort 8: 400mg/m2 (N=7) | Phase 2a Cohort 9: 400mg/m2 (N=17)
pneumonia (Infections and infestations) | 1 (1) | 2 (4) | 2 (3) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 6 (9) | 3 (3)
cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hemorrhage intracranial (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
histiocytosis hematophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
enterocolitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
enterobacter bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ecthyma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
escherichia bacteremia/sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
enterococcla infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: 50mg/m2 (N=3) | Phase 1 Cohort 2: 100mg/m2 (N=3) | Phase 1 Cohort 3: 200mg/m2 (N=4) | Phase 1 Cohort 4: 300mg/m2 (N=4) | Phase 1 Cohort 5: 400mg/m2 (N=7) | Phase 1 Cohort 6: 500mg/m2 (N=5) | Phase 1 Cohort 7: 400mg/m2 (N=5) | Phase 1 Cohort 8: 400mg/m2 (N=7) | Phase 2a Cohort 9: 400mg/m2 (N=17)
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0
atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 3
constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 4 | 2 | 1 | 1 | 0
diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 5 | 1 | 1 | 2 | 5
nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 5 | 1 | 1 | 3 | 7
stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 5
vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0
fatigue (General disorders) | 3 | 2 | 2 | 2 | 1 | 1 | 0 | 2 | 3
non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
edema peripheral (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4 | 0
pyrexia (General disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 4 | 0
alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0
blood bilirubin increased (Investigations) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0
platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
decreased appetitie (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 4 | 1 | 1 | 4 | 0
hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 3
hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 4 | 1 | 0 | 3 | 0
hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 3 | 3
hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 3 | 0
hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0
dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 4
confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 3
delirium (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 2 | 0 | 1 | 2 | 3
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 3 | 1 | 6
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02193958/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02193958/SAP_001.pdf